CLINICAL TRIAL: NCT01676519
Title: Impact of Critical Limb Ischemia on Long Term Cardiac Mortality in Diabetic Patients Undergoing Percutaneous Coronary Revascularization
Status: Completed | Type: Observational
Sponsor: Ospedale San Donato (Other)
Responsible Party: Principal Investigator, Leonardo Bolognese, MD, Director, Ospedale San Donato
Other Study IDs: Arezzo007
Record Dates: First submitted 2012-08-23; First posted 2012-08-31 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PCI: diabetic patients undergoing percutaneous coronary intervention
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI — percutaneous coronary intervention

SUMMARY:
Prospective cohort study of consecutive diabetic patients undergoing percutaneous coronary intervention (PCI) in whom development of critical limb ischemia was prospectively assessed by a dedicated diabetic foot clinic. Cardiac mortality at 4-year follow-up was the primary endpoint of the study.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus
* need for coronary revascularization
* age > 18 years

Exclusion Criteria:

* clinical contraindications to prolonged double antiplatelet therapy
* life expectancy < 1 year
* lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive diabetic patients undergoing percutaneous coronary intervention
Sampling Method: Probability Sample
Enrollment: 764 (Actual)
Dates: Start 2002-07; Primary Completion 2007-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
cardiac mortality rate | 4-year follow-up
  incidence of cardiac death

SECONDARY OUTCOMES:
major adverse cardiac event rate | 4-year follow-up
  incidence of major adverse cardiac events (cardiac death, myocardial infarction, target lesion revascularization)

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Department, Ospedale S.Donato, Arezzo, AR, Italy

REFERENCES:
- [Derived] Liistro F, Angioli P, Grotti S, Brandini R, Porto I, Ricci L, Tacconi D, Ducci K, Falsini G, Bellandi G, Bolognese L. Impact of critical limb ischemia on long-term cardiac mortality in diabetic patients undergoing percutaneous coronary revascularization. Diabetes Care. 2013 Jun;36(6):1495-500. doi: 10.2337/dc12-1603. Epub 2013 Jan 22. PMID 23340882